CLINICAL TRIAL: NCT06203678
Title: Investigation of the Effectiveness of Cervical Kinesio Taping Taping Application on Headache Symptoms in Migraine.
Brief Title: The Effectiveness of Cervical Kinesio Taping in Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-3
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Migraine; Kinesio Taping
Keywords: Migraine; Kinesio taping; Headache; Neck pain
MeSH Terms: conditions — Migraine Disorders; Headache; Neck Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio taping+exercise (Active Comparator): Kinesio taping will be applied to the bilateral upper trapezius and sternocleidomastoid muscles by an experienced practitioner, once a week for 4 weeks.
  Cervical stretching and strengthening exercises home program
  Interventions: Other: Kinesio taping; Other: Exercise
- Sham taping+exercise (Placebo Comparator): Sham taping will be applied to the bilateral upper trapezius and sternocleidomastoid muscles once a week for 4 weeks, using patch tape of the same color as kinesio tape.
  Cervical stretching and strengthening exercises home program
  Interventions: Other: Exercise; Other: Sham taping
- Exercise (Other): Cervical stretching and strengthening exercises home program
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Kinesio taping — therapeutic tape application
  Arms: Kinesio taping+exercise
Other: Exercise — Cervical stretching and strengthening exercises home program
Other: Sham taping — patch tape application
  Arms: Sham taping+exercise

SUMMARY:
Migraine is a common episodic headache disorder accompanied by neurological, gastrointestinal and autonomic changes.Migraine symptoms have a wide range, neck pain is seen in most migraine attacks, and accompanying neck pain is considered one of the important factors that increase migraine-related disability. It has been shown that various physical therapy methods applied to migraine patients with cervical myofascial pain reduce migraine pain and analgesic needs. One of the methods used in myofascial pain syndrome is kinesio taping and the effectiveness of cervical area applications has been shown in different studies.In this study, it was planned to examine the effect of kinesio taping applied to cervical trigger points on migraine symptoms in migraine patients.

DETAILED DESCRIPTION:
The annual prevalence of migraine is approximately 15% and it is the second most common neurological disease worldwide. Migraine symptoms have a wide range, neck pain is seen in most migraine attacks, and accompanying neck pain is considered one of the important factors that increase migraine-related disability. In myofascial pain syndrome, active trigger points are considered as the source of pain and the treatment goal is to relax and inhibit these trigger points. It has been shown that various physical therapy methods applied to migraine patients with cervical myofascial pain reduce migraine pain and analgesic needs. In a study conducted with forty migraine patients, a significant decrease in headache parameters was reported with dry needling applied to the sternocleidomastoid muscle immediately after the procedure and at 1-month follow-up. Similarly, in migraine patients who received local anesthetic injection and topical analgesic treatment for cervical myofascial pain in addition to migraine prophylaxis, a decrease in attack frequency, severity and analgesic need was found compared to the control group.Kinesio taping is one of the most preferred conservative treatments for pain originating from the musculoskeletal system, and it is suggested that it provides an increase in blood and lymphatic flow by applying tension force on the skin with its elastic structure, and provides muscle relaxation with proprioceptive stimulation. In this study, it was planned to examine the effect of kinesiology taping applied to the cervical region on migraine symptoms in migraine patients.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of migraine without aura for at least 1 year according to the International Classification of Headache Disorders criteria
* Being under migraine prophylactic treatment
* Being between the ages of 18-65
* Physical examination reveals a cervical (trapezoidal and SCM) myofascial trigger point with a spreading pattern overlapping the migraine pain area.
* Being literate
* Agreeing to participate in the study

Exclusion Criteria:

* History of neck trauma, cervical radiculopathy and previous cervical surgery
* Physical therapy, injection and manipulation to the cervical area in the last 3 months
* History of fibromyalgia, active cancer, systemic inflammatory disease and infection
* Pregnancy
* Being <18 and >65 years old
* Being illiterate

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female patients diagnosed with migraine
Enrollment: 18 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
headache index (HI) | 3 months
  HI is calculate as mean migraine days per month (30 days) × mean migraine duration (h/day) × mean intensity (0-10 numeric rating scale).

SECONDARY OUTCOMES:
Migraine day | 3 months
  A migraine day is defined as the day on which migraine with or without aura or possible migraine occurs.
number of migraine days per month (30 days/month) | 3 months
  number of migraine days per month (30 days/month)
migraine duration | 3 months
  Migraine pain duration (hour)
numeric rating scale | 3 months
  The numeric rating scale (NRS) is a validated subjective measure for pain, scored in the 0-10 range (0:no pain; 10: worst pain).
The Migraine Disability Assessment Test | 3 months
  This scale is used to evaluate headache-related disability in migraine patients. Accordingly, 0-5 points; Stage 1, 6-10 points; Stage 2; 11-20 points; Stage 3; Scores of 21 points and above are classified as Stage 4, and as the stage increases, the severity of disability increases.
hospital anxiety and depression scale | 3 months
  This scale is used to screen for anxiety and depression in individuals with physical illnesses.The scale consists of a total of 14 questions, 7 of which are anxiety and 7 depression, to be answered on a four-point Likert scale. A score above 10 for anxiety and 7 points for depression is considered significant.
24-Hour Migraine Quality of Life Questionnaire (24-Hr MQoLQ) | 3 months
  A 24-Hour Migraine Quality of Life Questionnaire (24-Hr MQoLQ) is a scale to measure the decrease of quality of life of a person within the past 24 hours after suffering of an acute migraine and taking migraine medication.The scale consists of 15 Likert-type questions scored in the range of 0-5, with higher scores indicating more deterioration in quality of life.
Cervical range of motion | 3 months
  Cervical joint range of motion measurement with inclinometer (includes flexion, extension, lateral flexion and rotations)
Pressure pain threshold | 3 months
  Pain pressure threshold (PPT) is used to measure deep muscular tissue sensitivity. Algometer is used in the measurement and low values are interpreted in favor of increased sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Ata, Assoc.Prof, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Sultan Abdülhamid Han Training and Research Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
no data sharing planned

REFERENCES:
- [Result] Eigenbrodt AK, Ashina H, Khan S, Diener HC, Mitsikostas DD, Sinclair AJ, Pozo-Rosich P, Martelletti P, Ducros A, Lanteri-Minet M, Braschinsky M, Del Rio MS, Daniel O, Ozge A, Mammadbayli A, Arons M, Skorobogatykh K, Romanenko V, Terwindt GM, Paemeleire K, Sacco S, Reuter U, Lampl C, Schytz HW, Katsarava Z, Steiner TJ, Ashina M. Diagnosis and management of migraine in ten steps. Nat Rev Neurol. 2021 Aug;17(8):501-514. doi: 10.1038/s41582-021-00509-5. Epub 2021 Jun 18. PMID 34145431
- [Result] Gandolfi M, Geroin C, Vale N, Marchioretto F, Turrina A, Dimitrova E, Tamburin S, Serina A, Castellazzi P, Meschieri A, Ricard F, Saltuari L, Picelli A, Smania N. Does myofascial and trigger point treatment reduce pain and analgesic intake in patients undergoing onabotulinumtoxinA injection due to chronic intractable migraine? Eur J Phys Rehabil Med. 2018 Feb;54(1):1-12. doi: 10.23736/S1973-9087.17.04568-3. Epub 2017 Jul 27. PMID 28750504
- [Result] Rezaeian T, Ahmadi M, Mosallanezhad Z, Nourbakhsh MR. The impact of myofascial release and stretching techniques on the clinical outcomes of migraine headache: A randomized controlled trial. J Res Med Sci. 2021 Jul 31;26:45. doi: 10.4103/jrms.JRMS_745_18. eCollection 2021. PMID 34484377
- [Result] Rezaeian T, Mosallanezhad Z, Nourbakhsh MR, Noroozi M, Sajedi F. Effects of Dry Needling Technique Into Trigger Points of the Sternocleidomastoid Muscle in Migraine Headache: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2020 Dec;99(12):1129-1137. doi: 10.1097/PHM.0000000000001504. PMID 32544109
- [Result] Affaitati G, Costantini R, Tana C, Lapenna D, Schiavone C, Cipollone F, Giamberardino MA. Effects of topical vs injection treatment of cervical myofascial trigger points on headache symptoms in migraine patients: a retrospective analysis. J Headache Pain. 2018 Nov 8;19(1):104. doi: 10.1186/s10194-018-0934-3. PMID 30409108
- [Result] Unlu Ozkan F, Soylu Boy FN, Erdem Kilic S, Geler Kulcu D, Bicer Ozdemir G, Cagliyan Hartevioglu H, Akpinar P, Aktas I. Clinical and radiological outcomes of kinesiotaping in patients with chronic neck pain: A double-blinded, randomized, placebo-controlled study. Turk J Phys Med Rehabil. 2020 Nov 9;66(4):459-467. doi: 10.5606/tftrd.2020.5632. eCollection 2020 Dec. PMID 33364567